CLINICAL TRIAL: NCT04181996
Title: The Canadian Study of Arterial Inflammation in Patients With Diabetes and Recent Vascular Events: EvaluatioN of Colchicine Effectiveness (CADENCE)
Brief Title: Canadian Study of Arterial Inflammation in Patients With Diabetes and Vascular Events: EvaluatioN of Colchicine
Acronym: CADENCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB # - 20190355-01H CRRF:1443
Record Dates: First submitted 2019-11-19; First posted 2019-12-02 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Inflammation; Diabetes
Keywords: Imaging, PET, inflammation, Biomarkers, Colchicine
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Inflammation; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind Placebo controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo: Sugar pill manufactured to mimic colchicine 0.6 mg capsule. Placebo to be taken once a day.
  Interventions: Drug: Placebo oral capsule
- Colchicine (Experimental): Colchicine: 0.6 mg colchicine capsule to be taken once a day.
  Interventions: Drug: Colchicine Oral Product

INTERVENTIONS:
Drug: Colchicine Oral Product — Patients will be randomized to receive either placebo or colchicine
  Arms: Colchicine
Drug: Placebo oral capsule — Patents will be randomized to receive either placebo or colchicine
  Arms: Placebo

SUMMARY:
Cardiovascular Disease (CVD) is a leading cause of death in the developed world. Atherosclerosis causes plaques in the blood vessels and is a common form of CVD. Inflammation is now recognized as a major cause of atherosclerosis. Therapies that target inflammation are being examined as a potential treatment option. Imaging to detect inflammation may be a solution to understand mechanisms and to optimize patient selection and outcomes for these drugs. Fluorodeoxyglucose (FDG) PET imaging can detect inflammation in the plaque and identify patients vulnerable to plaque rupture which cause events such as myocardial infarctions (MI) and strokes. The primary objective of this proposal(CADENCE) is to determine if the drug colchicine has an effect on plaque inflammation in patients at high risk for events (patients with diabetes or pre-diabetes and recent myocardial infarction, stroke or transient ischemic attacks (TIAs)). This mechanistic and proof-of-concept study will set the stage for future studies that will determine if inflammation imaging can be integrated into clinical practice to personalize decisions for anti-inflammation therapies.

DETAILED DESCRIPTION:
Inflammation is a key to atherosclerosis and its serious effects (MI, stroke) and represents a potentially transformative therapeutic target. Several recent trials have revealed potential outcome benefit in patients with cardiovascular disease who are treated with anti-inflammatory therapy. The LoDoCo trial showed a reduction in cardiovascular events in patients with known coronary artery disease who were treated with colchicine (1). Although the LoDoCo trial did show outcome benefit, and in fact reduced the number of acute coronary syndromes in the treatment group, colchicine's mechanism of action at the level of the atherosclerotic plaque in patients remains unknown. The COLCOT trial was recently published which further demonstrated the potential benefit of anti-inflammatory therapy with colchicine. Compared with placebo, colchicine significantly reduced the risk of cardiovascular events for patients who recently experienced a myocardial infarction (2). It is not clear at the present time whether colchicine mainly reduces the systemic inflammatory milieu, thus reducing the likelihood of plaque progression and new lesion formation; or whether it has a direct effect on local "hot" inflammatory cell activity, thus pacifying the inflammatory plaque to reduce events. Insight into colchicine's mechanism of action may help identify the most suitable patients for this novel approach.

Inflammation imaging may represent a solution. 18F-fluorodeoxyglucose (FDG) PET-CT imaging can define plaque inflammation and identify patients and plaques vulnerable to rupture and events. Improved FDG uptake occurs with therapies that effectively reduced vascular events but not with therapies with no outcome benefit. It is provocative to consider inflammation imaging strategies that may positively impact therapy decisions to yield better patient selection and outcomes.

The long term goal of this research is to determine the pathobiological effect of colchicine on plaque inflammation and determine if inflammation imaging can be integrated into clinical assessment to personalize decisions for anti-inflammation therapies. As the first step for this goal, the investigators propose The CADENCE study is the first step towards this goal; it is a mechanistic and proof-of-concept study that will be the basis for a future 2nd phase definitive RCT integrating inflammation imaging and biomarker strategies.

The Primary Objective is to determine the pathobiological effect of the medication colchicine compared to placebo, on plaque inflammation (measured by 18F-fluordeoxyglucose (FDG) PET/CT at baseline and 6 months) in the carotid arteries and thoracic aorta in high-risk patients with diabetes or pre-diabetes and recent vascular events (ACS/MI, TIA, stroke) to investigate whether its mechanism of action is primarily systemic or local at the plaque level. FDG PET/CT has been demonstrated to offer a pragmatic method to assess inflammation in the aorta.1 Several studies confirm that therapies that reduce aortic FDG uptake mirror clinical efficacy..

Secondary Objectives are to determine: a) whether baseline inflammation imaging (FDG PET/CT) and/or inflammation biomarker (hs-CRP) levels can identify the patients most likely to have a positive response to colchicine measured by the change in FDG uptake over 6 months; b) the relationship of the inflammation response on FDG PET/CT to hs-CRP at baseline and over the 6-month time-frame.

Exploratory Objectives are to determine: a) if there are regional differences (i.e. carotid or aorta) in response to colchicine in patients with recent coronary (ACS/MI) versus those with recent cerebral events (TIA, stroke); b) if other systemic inflammation biomarkers (e.g, IL-6, IL-1β, TNF-α, MCP-1, others) also predict the response to colchicine; c) the relationship of inflammation on FDG PET/CT to: i) systemic inflammation biomarkers; ii) monocyte activation; d) treatment effect on clinical outcomes such as major adverse CV events and all-cause mortality; and e) the effect on quality of life outcomes.

Methods:

In CADENCE patients with T2DM or pre-diabetes and a recent NonSTEMI, STEMI, stroke or TIA will be recruited to one of 2 arms: colchicine 0.6 mg daily; or placebo. At baseline and 6 months: patients will have FDG PET-CT of carotids and aorta; at 0, 3 and 6 months: clinical evaluation and blood sampling for inflammation biomarkers (eg hsCRP, IL-6, IL-1β, TNF-α, MCP-1). The primary endpoint will be the change in inflammation over 6 months measured as FDG tissue to blood ratio (TBR).

Expected Outcomes:

It is expected that colchicine will reduce arterial inflammation measured using FDG PET/CT and reduce biomarkers of systemic inflammation. This would validate that colchicine's mechanism of action is more than a systemic effect but also a local action at the level of the vessel wall and plaque. This would further identify arterial inflammation on imaging as a potential novel therapeutic target for those at high risk of CV events. Such proof-of-concept data would support a definitive RCT to evaluate and define the potential for new biomarker-imaging strategies to direct decisions for novel anti-inflammation therapies in this population.

Current therapies focus on lesion stenosis or ischemia with conflicting results. Use of inflammation imaging to direct proven treatments would be a bold practice-changing paradigm shift.

ELIGIBILITY:
Inclusion Criteria:

Patients who have:

1. Type 2 Diabetes (on diet, oral hypo-glycemic agents and/or insulin) or pre-diabetes (defined by Diabetes Canada as HbA1C=6.0-6.45% or increased fasting blood sugar (FBS) (6.1-6.9 mmol/L) or impaired glucose tolerance);
2. suffered a recent cardiovascular event (≤120 days post ACS (i.e. STEMI or nonSTEMI) or TIA/stroke with associated large vessel atherosclerotic disease confirmed on US, CT or MRI;
3. stable symptoms and hemodynamics;
4. age ≥18 years;
5. given informed consent. Standard definitions will be used for STEMI, NSTEMI, and for ischemic stroke confirmed by CT or MRI and TIA confirmed by a neurologist.

Exclusion Criteria:

Patients who have

1. planned revascularization of infarct or stroke related artery more than 120 days after the qualifying/index event;
2. a recent CV event likely to have been embolic in the opinion of the neurologist or cardiologist;
3. recent CV event likely to have been secondary to myocardial infarction with non-obstructive coronary arteries (MINOCA) in the opinion of the cardiologist;
4. severe LV dysfunction (EF<30%);
5. severe valve disease requiring intervention;
6. decompensated heart failure;
7. active infection (e.g. pneumonia, active skin infections, and on antibiotics);
8. chronic diarrhea;
9. immune compromise (e.g. recurrent infection);
10. history of cancer within the last 3 years (other than a successfully treated cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix).
11. active inflammatory conditions (e.g. rheumatoid arthritis, chronic inflammatory bowel disease, SLE, systemic anti-inflammatory therapy (e.g. prednisone, methotrexate));
12. pregnancy (all women of child bearing potential will have a negative BHCG test;
13. breastfeeding;
14. Women of childbearing potential who refuse to use two forms of contraception (this includes at least one form of highly effective and one effective method of contraception) throughout the study OR men capable of fathering a child who refuse to use contraception.
15. glomerular filtration rate (GFR) <50 ml/min/1.72m2
16. Use of potent p-glycoprotein inhibitors (i.e. systemic cyclosporine, clarithromycin, or systemic ketoconazole) or a strong CYP3A4 inhibitor (i.e. ritonavir, clarithromycin, or systemic ketoconazole);
17. Hemoglobin < 105(women) <110 (men) g/L; WBC < 3.0x 10(9)/L, platelet count< 110x 10(9)/L;
18. Patient with a history of cirrhosis, chronic active hepatitis or severe hepatic disease or with alanine aminotransferase (ALT) levels greater than 3 times the upper limit of normal.
19. unable to give informed consent;
20. TIA/Stroke patients with atrial fibrillation

Exclusion for CTA portion of the protocol:

Patients with dye allergy or those with GRF <60 will not undergo CTA but will have PET/CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-08-14 (Estimated); Study Completion 2025-08-14 (Estimated)

PRIMARY OUTCOMES:
6 month change in FDG uptake TBR (Tissue to Blood Ratio) in the MDS (Maximum Disease Segment) | 6 months
  The primary endpoint will be the change over 6 months in the FDG uptake TBR (Tissue-to-blood ratio) as a marker of arterial plaque inflammation in the maximum disease segment (MDS)(the segment with the highest TBR at baseline) in any vasculature imaged whether it be left or right carotid or aorta.

SECONDARY OUTCOMES:
6 month change in FDG uptake TBR (Tissue to Blood Ratio) in the MDS of each vascular region: aorta, left and right carotid. | 6 months
  6 month change in FDG uptake TBR (Tissue to Blood Ratio) in the MDS of each vascular region: aorta, left and right carotid.
6 month change in FDG uptake SUV (standard uptake value) in the MDS of each vascular region: aorta, left and right carotid. | 6 months
  6 month change in FDG uptake SUV (standard uptake value) in the MDS of each vascular region: aorta, left and right carotid.
Levels of high-sensitivity C-Reactive Protein (hs-CRP) (mg/ml) and its change | 6 months
  Levels of high-sensitivity C-Reactive Protein (hs-CRP) (mg/ml) and its change
Levels of Interleukin-6 (IL-6) (pg/ml) and its change. | 6 months
  Levels of Interleukin-6 (IL-6) (pg/ml) and its change.

OTHER OUTCOMES:
Exploratory outcomes - Plasma levels of cytokines (pg/ml) | 6 months
  Plasma levels of other cytokines (pg/ml)
Exploratory outcomes - Levels of activated monocytes | 6 months
  Levels of activated monocytes
Exploratory outcomes - plasma levels of inflammation biomarkers | 6 months
  Plasma levels of inflammation biomarkers
Exploratory outcomes - MACE | 6 months
  MACE (multiple adverse CV events (ACS/MI, TIA, stroke, CV death))
Exploratory outcomes - non CV death | 6 months
  non-cardiovascular death
Exploratory outcomes - treatment effect on clinical outcomes such as major adverse CV events and all-cause mortality | 6 months
  Exploratory outcomes - treatment effect on clinical outcomes such as major adverse CV events and all-cause mortality
Exploratory outcomes - the effect on quality of life outcomes | 6 months
  Exploratory outcomes - the effect on quality of life outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Boczar, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - University of Ottawa Heart Institute, Ottawa, Ontario

REFERENCES:
- [Background] Nidorf SM, Eikelboom JW, Budgeon CA, Thompson PL. Low-dose colchicine for secondary prevention of cardiovascular disease. J Am Coll Cardiol. 2013 Jan 29;61(4):404-410. doi: 10.1016/j.jacc.2012.10.027. Epub 2012 Dec 19. PMID 23265346
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Derived] Boczar KE, Shin S, deKemp RA, Dowlatshahi D, Tavoosi A, Wiefels C, Liu P, Lochnan H, MacPherson PA, Chong AY, Torres C, Leung E, Tawakol A, Ahmadi A, Garrard L, Lefebvre C, Kelly C, MacPhee P, Tilokee E, Raggi P, Wells GA, Beanlands R. The Canadian Study of Arterial Inflammation in Patients with Diabetes and Recent Vascular Events, Evaluation of Colchicine Effectiveness (CADENCE): protocol for a randomised, double-blind, placebo-controlled trial. BMJ Open. 2023 Nov 10;13(11):e074463. doi: 10.1136/bmjopen-2023-074463. PMID 37949621